CLINICAL TRIAL: NCT03870698
Title: Comparison of Perioperative Outcomes Between Laparoscopic and Open Pylorus Preserving Pancreaticoduodenectomy in Periampullary Tumors: Randomized Controlled Study
Brief Title: Comparison of Functional Recovery Between Laparoscopic and Open Pancreaticoduodenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Severance Hospital (Other); Samsung Medical Center (Other); Hallym University Medical Center (Other)
Responsible Party: Principal Investigator, Song Cheol Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CORLAPPD_01
Record Dates: First submitted 2019-03-06; First posted 2019-03-12 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Functional Recovery; Laparoscopy; Periampullary Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic group (Experimental): The patients who underwent laparoscopic procedures for periampullary tumors
  Interventions: Procedure: Laparoscopic group
- Open group (No Intervention): The patients who underwent open procedures for periampullary tumors

INTERVENTIONS:
Procedure: Laparoscopic group — The patients in laparoscopic group will underwent pylorus preserving pancreaticoduodenectomy in laparoscopic manners.
  Arms: Laparoscopic group

SUMMARY:
Laparoscopic surgery has not changed much in safety compared with open surgery through many existing studies, and has become a procedure to help patients' recovery.

Recently, laparoscopic surgery has been actively performed for pancreaticoduodenectomy, one of the most complicated procedures in intraperitoneal surgery.

the investigators will perform a prospective study to establish a higher level of evidence for the efficacy and safety of laparoscopic pancreaticoduodenectomy.

The purpose of this study was to compare the short-term clinical outcomes including the functional recovery after surgery, complications and confirm that laparoscopic pancreaticoduodenectomy is safe and appropriate. This study includes an interim analysis and can be terminated early by analysis at the completion of 50% of planned patients.

DETAILED DESCRIPTION:
* Pancreatoduodenectomy is a standard procedure for periampullary disease of the duodenum (pancreatic cancer, biliary pancreatic cancer, bile duct cancer, etc.) and is a very extensive and complicated operation for partial resection of the pancreas, duodenum, bile duct, gallbladder and occasionally stomach. In addition, anastomotic anastomoses are considered to be one of the most complicated surgeries among intraperitoneal procedures, even in open surgery. Laparoscopic surgery has been advancing rapidly with the development of the technique of laparoscopic surgery. In recent years, Pancreatoduodenectomy has been actively attempting laparoscopic surgery centering on large organs. As a result, large incision and abdominal wall traction can be avoided. Common advantages include postoperative pain relief, rapid recovery of bowel movements, fewer days of hospitalization, and a quick return to daily life. In addition, recently reported meta-analysis has shown that laparoscopic Pancreatoduodenectomy has a significantly lower bleeding volume and duration of hospitalization compared to open surgery.
* This study was aimed to compared functional recovery between open and laparoscopic PD in 3 tertiary referral centers in Korea. The investigators will measure functional recovery .
* A case of pancreaticoduodenectomy with benign tumor in the pancreas will be included. The expected number of patients is 252. The laparoscopic surgery was performed in the experimental group and the open surgery was performed in the control group. When achieving 50% of the planned target group, the interim analysis will decide whether to continue the study.

This clinical study is a randomized prospective comparative study of the outcome of laparoscopic and open Pancreatoduodenectomy, and the research hypothesis is as follows.

* Nursing Hypothesis: There is no difference in the functional recovery between patients who underwent laparoscopic pancreaticoduodenectomy and patients who underwent open surgery.
* Alternative Hypothesis: Based on the results of the same operation of the existing institution, the average functional recovery for open pancreaticoduodenectomy is estimated to be 14 days, and the functional recovery for laparoscopic pancreaticoduodenectomy is reduced by 20%.

The random assignment of this study is assigned according to the order of assignment in the planning stage of the study as a block randomization scheme with appropriate block size set.

* Plan for recruitment of research subjects All patients who underwent pancreaticoduodenectomy for the pancreas or peripapillary lesion were selected and selected as subjects after explaining the study and accepting consent.
* Operative methods Both patients underwent conventional pancreaticoduodenectomy or pyloric preservation pancreaticoduodenectomy. In the control group, the midline incision was performed and the operation was performed by the laparotomy. In the experimental group, laparoscopic surgery was performed using 5-6 trocars. Laparoscopy and laparotomy are performed through the same surgical procedure and the procedure is as follows. Kocher maneuver is performed to mobilize the duodenum.

Omentectomy is performed and the gastrocolic truck is identified and ligated. The stomach or duodenum is cut off using an automatic stapler. A cholecystectomy is performed. The bile duct is cut and the frozen section is checked to confirm whether the tumor is invaded. The hepatic and hepatic arteries are dissected and the surrounding lymph nodes are dissected. The gastroduodenal artery is detached and ligated. The pancreas is cut from the pancreas neck, and the tumor is examined by freezing biopsy. The proximal plant is dissected and cut, and the pancreas uncinate process is released from the superior mesenteric artery and vein. Pancreaticojejunal anastomosis, hepaticojejunal anastomosis, gastrojejunal or duodenojejunal anastomosis are performed. In this case, anastomosis is performed by the method used by each institution.

Indications for open conversion

* In a situation where the safety of the patient is threatened, it is possible to switch to the opener at any time under the judgment of the researcher.
* Vascular involvement of the superior mesenteric vein, superior mesenteric artery, and hepatic artery is suspected and the operation is difficult to perform.
* The operation is difficult due to severe pancreatitis
* Laparoscopic treatment is difficult if there is bleeding

Patient management after surgery.

* 1 day after surgery: Removal of blood and nasogastric tube after surgery, water intake, early gait, cytokine check
* 2 days after surgery: initiation or death, cytokine check
* 3 days after surgery: intravenous patient controlled analgesia removal, after 3 days, considering drain amylase and drain volume can be removed. Check functional recovery daily after 3 days
* 5 days after surgery: Perform computed tomography.
* 7 days after surgery: If the patient is a malignant tumor, the tumor marker will be collected. Cytokine check

ELIGIBILITY:
Inclusion Criteria:

* Age: 19 to 80 years
* Performance: Eastern Cooperative Oncology Group (ECOG) 0-2
* The preoperative examination showed that the lesion could not be invaded by major blood vessels.
* No distant metastasis
* Bone marrow function: white blood cell (WBC) at least 3,000 / mm3, Platelet count at least 100,000 / mm3
* Kidney function: Creatinine no greater than 1.5 times upper limit of normal.
* Patients who consented to and signed the consent

Exclusion Criteria:

* Severe obesity (BMI> 30)
* Those with active or uncontrolled infections
* Those with severe psychiatric / neurological disorders
* Alcohol or other drug addicts
* Patients included in other clinical studies that may affect this study
* Patients who cannot follow the directions of the researcher
* Those with uncontrolled heart disease
* Patients with moderate or severe comorbidities who are thought to have an impact on quality of life or nutritional status (cirrhosis, chronic kidney failure, heart failure, etc.)
* Pelvic tumor, benign tumor, malignant tumor in other organs
* Patients who received prior chemotherapy
* In addition to the planned PD patients who require resection of other major abdominal organs (such as gastrectomy, colonic resection and portal / upper mesenteric vascular resection, more than standard PD)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Time to functional recovery after surgery | up to 1 months
  It is defined that functional recovery is achieved if all of the following are satisfied.
  1. Pain can be controlled by oral or patch analgesic without intravenous analgesics. * 2. Free walking (modified enhanced recovery after surgery mobility scale 5/5) ** 3. Free diet is available (more than 1/2 of the dietary intake) 4. No evidence of infection (body temperature <38.5 degrees, C-reactive protein (CRP) 15 mg / dL, no complicated fluid collection on postoperative computed tomography 5. There should be no intravenous injection .

SECONDARY OUTCOMES:
Numbers of Hospital stay | up to 2 months
  It is defined that discharge day after surgery
Minutes of operation time | Up to 1 day after surgery
  It mean time from anesthesia to end of surgery
amount of estimated blood loss | up to 1 day after surgery
  It means amount of bleeding during surgery
Severity of postoperative pain | Up to 3 days
  It refers to the degree of pain measured during 2 days after surgery
postoperative complications | up to 2 months
  It means all kinds of complications after surgery
Numbers of complete resection in pathological results | Up to 2weeks
  It means no remnant tumor in pathologic results
level of serum cytokine | Up to 1 week
  It means value of serum cytokine, which was collected after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Song-Cheol Kim, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yoon YS, Lee W, Kang CM, Hong T, Shin SH, Lee JW, Hwang DW, Song KB, Kwon JW, Sung MK, Shim IK, Lee JB, Kim SC; for Korean Study Group on Minimally Invasive Pancreatic Surgery (K-MIPS). Laparoscopic versus open pancreatoduodenectomy for periampullary tumors: a randomized clinical trial. Int J Surg. 2024 Nov 1;110(11):7011-7019. doi: 10.1097/JS9.0000000000002035. PMID 39172725